CLINICAL TRIAL: NCT06433895
Title: Efficacy of Manual Therapy in the Treatment of Somatic Tinnitus: A Randomised Controlled Trial
Brief Title: Efficacy of Manual Therapy in the Treatment of Somatic Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tuğba Atan, MD, Assoc. Prof., Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-21-1003
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-06

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual therapy + Exercise group (Experimental): Both groups will be instructed in the performance of isometric and strengthening exercises for the cervical region, which are provided to patients with cervical pain and limitation as a home programme for a six-week period. Additionally, patients in the manual therapy group will receive manual therapy on a weekly basis for a total of six sessions.
  Interventions: Other: Manual Therapy; Other: Exercise
- Exercise group (Active Comparator): Both groups will be instructed in the performance of isometric and strengthening exercises for the cervical region, which are provided to patients with cervical pain and limitation as a home programme for a six-week period.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Manual Therapy — Manual Therapy
  Arms: Manual therapy + Exercise group
Other: Exercise — Isometric and strengthening exercises for the cervical region, which are provided to patients with cervical pain and limitation

SUMMARY:
Somatic tinnitus is an unpleasant perception of sound that occurs in the absence of any external acoustic stimulus. Despite the correct diagnosis of somatic tinnitus, there is currently no specific treatment. The hypothesis of this study is that the application of manual therapy to the cervical region will help to treat tinnitus in patients. This study aims to investigate the effectiveness of manual therapy in the treatment of somatic tinnitus of cervicogenic origin.

DETAILED DESCRIPTION:
Somatic tinnitus is an unpleasant perception of sound that occurs in the absence of any external acoustic stimulus. It results from complex interactions between the somatosensory and auditory systems, which involve the musculoskeletal system rather than the ear. The temporomandibular joint, craniocervical junction, cervical vertebrae and neck and shoulder muscles, in particular the sternocleidomastoid (SCM) muscle, upper trapezius and levator scapula, are anatomical regions that can cause somatic tinnitus.

Despite the correct diagnosis of somatic tinnitus, there is currently no specific treatment. The hypothesis of this study is that the application of manual therapy to the cervical region will help to treat tinnitus in patients. This study aims to investigate the effectiveness of manual therapy in the treatment of somatic tinnitus of cervicogenic origin.

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥ 18 and ≤ 65 years Patients fulfilling the clinical criteria4 defined for sevichogenic somatic tinnitus

1. Neck pain
2. Cervical joint range of motion limitation (especially rotation)
3. Modulation of tinnitus in relation to head and neck movements and posture
4. Tenderness in the cervico-occipital muscles Patients reporting cervical pain between >2 and <7 on a visual analogue scale (VAS) on most days of the last month Patients with stable medical and psychological status Patients willing to participate in the study

Exclusion Criteria:

Objective tinnitus Subjective tinnitus with hearing loss Meniere's disease History of vertigo Middle ear pathologies History of intracranial pathology History of whiplash injury History of cervical spinal surgery History of active infection, malignancy, inflammatory rheumatic disease or fibromyalgia Pregnancy Patients who have undergone any exercise or physiotherapy programme for the cervical region in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-05-25 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Tinnitus (VAS-tinnitus) | baseline- 6 week
  The severity of tinnitus will be graded using a 10 cm visual analogue scale (VAS, 0-10 cm; 0 means no tinnitus, 10 means extremely severe tinnitus).

SECONDARY OUTCOMES:
Visual Analogue Scale for cervical pain (VAS-Cervical) | baseline- 6 week
  Pain intensity will be assessed with the visual analogue scale (0-10mm), which has proven validity and reliability for measuring musculoskeletal pain.
Tinnitus Handicap Index (THI) | baseline- 6 week
  The THI contains a total of 25 items with functional (11 items), emotional (9 items) and catastrophic (5 items) subscales. Each item is rated 0 (not affected), 2 (sometimes affected) or 4 (always affected). The total score ranges from 0 to 100, with higher scores indicating higher levels of disability of perceived tinnitus.
Neck disability index (NDI) | baseline- 6 week
  The NDI is designed to assess self-reported neck functional status. The questionnaire consists of 10 items related to pain, activities of daily living, weight lifting, reading, headache, concentration, working status, driving, sleep and recreation and is rated on a 6-point Likert scale ranging from 0 (no disability) to 50 (major disability). Higher scores represent greater disability. The NDI has been found to be reliable and valid for cervical disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Educiation and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No